CLINICAL TRIAL: NCT04916405
Title: Standardized Management of Pregnancy Weight of Twin Pregnancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Caixia Liu (Other)
Responsible Party: Sponsor-Investigator, Caixia Liu, Clinical Professor, Shengjing Hospital
Organization: Shengjing Hospital (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: PWOTP
Record Dates: First submitted 2021-05-26; First posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Pregnancy Weight of Twin Pregnancy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Standardized management of pregnancy weight of twin pregnancy — Standardized management of pregnancy weight of twin pregnancy

SUMMARY:
There are few studies on the optimal value of pregnancy weight gain for twin pregnancy in China.At present, China has not put forward guidelines for the appropriate value of weight gain in twin pregnancy, and the lack of standards for weight gain during pregnancy in clinical application or disease prevention and control seriously restricts the health management of pregnant women.In order to effectively control a series of adverse consequences caused by improper weight gain of women during twin pregnancy, it is urgent to establish the appropriate value of weight gain during twin pregnancy, which will also fill the gap in this field in China.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years
* Twin pregnancy
* pregnancy weeks ≤ 6 weeks

Exclusion Criteria:

* adverse pregnancy history
* kidney disease

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Weight gain of women during twin pregnancy | 1 year

IPD SHARING:
Plan to Share IPD: Undecided